CLINICAL TRIAL: NCT05127408
Title: Endoscopic Sutures for Gastrointestinal Tract Disorders: A Prospective Multicenter Registry
Brief Title: Gastrointestinal Tract Disorders: A Prospective Multicenter Registry
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 021.GID.2019.D
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Endoscopic Suturing; GI Tract Disorders; Gastrointestinal Disorders
Keywords: Sutures; gi
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Interventional Endoscopy — correct defects of the gastrointestinal tract.
  Other Names: Apollo Endosurgery OverStitch™ Endoscopic Suture System (ESS) (or Endo Stitch™ , the SILS™ Stitch)

SUMMARY:
The purpose of this prospective registry is to assess long-term data on efficacy, safety and clinical outcome of endoscopic placement of suture(s) and approximation of soft tissue within the gastrointestinal tract for various GI tract disorders. Currently, lack enough data evaluate and verify technical feasibility, clinical success and safety of endoscopic suturing in specific gastrointestinal disorders.1-16 Evaluation of these factors would help us compare them to conventional treatment modalities; and consequently help us identify appropriate treatment techniques and improve clinical management of patients.

DETAILED DESCRIPTION:
This study is a prospective, observational, medical chart review for at least six standards of care visits up to 1 year after subject consents for study participation. There will be a retrospective chart review for patients who underwent endoscopic suturing procedures from October 2014 - April 2019. Those subjects will undergo no additional tests and procedures as part of this study. All data will be collected from patient's electronic health records (EHR) of the hospital In addition; a prospective chart review will be performed for patients who will undergo endoscopic suturing procedures from April 2019 to April 2021. All the subjects enrolled in prospective chart review will be first consented for their study participation. Subjects will undergo a clinically indicated endoscopic suturing procedure and standard of care follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has undergone clinically indicated and/or standard of care endoscopic suturing within the Gastrointestinal tract
* Above or equal to 18 years of age

Exclusion Criteria:

* Any patient who has not undergone endoscopic suturing within the gastrointestinal tract
* Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who has undergone clinically indicated and/or standard of care endoscopic suturing within the Gastrointestinal tract at Methodist Health System in Dallas.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Documentation of successful procedures. | October 2014 to April 2021
  Documentation of technical success (in terms of technical feasibility) Documentation of clinical success rates. Documentation of Safety: Number of subjects with Adverse Events; Type, frequency and intensity of adverse events

SECONDARY OUTCOMES:
Documentation of unsuccessful procedures. | October 2014 to April 2021
  Documentation of follow up adverse events and recurrence of initial GI disorder

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Kedia, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided